CLINICAL TRIAL: NCT03203005
Title: A Phase I/II Trial of IMA970A Plus CV8102 Following a Single Pre-vaccination Infusion of Cyclophosphamide in Patients With Very Early, Early and Intermediate Stage of Hepatocellular Carcinoma After Any Standard Treatments
Brief Title: IMA970A Plus CV8102 in Very Early, Early and Intermediate Stage Hepatocellular Carcinoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Immatics Biotechnologies GmbH (Industry); CureVac (Industry); European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HepaVac-101
Record Dates: First submitted 2017-06-13; First posted 2017-06-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMA970A plus CV8102 and Cyclophosphamide (Experimental): Investigational treatment with IMA970A, CV8102, Cyclophosphamide
  Interventions: Drug: IMA970A plus CV8102 and Cyclophosphamide

INTERVENTIONS:
Drug: IMA970A plus CV8102 and Cyclophosphamide — Study treatment starts with a single intravenous infusion of 300mg/m2 Cyclophosphamide.
  Three days later patients start vaccination therapy with IMA970A plus CV8102 Each vaccination consists of a dose of 6.80 milligrams (mg) IMA970A (containing approx. 400 micrograms [µg] of each individual peptide) followed by a dose of 50 µg CV8102. First IMA970A is injected intradermally (i.d.) and about 10 minutes later CV8102 is injected i.d. at the same vaccination site in close proximity. Patients will receive 4 vaccinations at weekly intervals followed by 5 vaccinations at 3-weekly intervals for a total duration of about 4.5 months.
  Other Names: Cyclophosphamide Injection 1 g

SUMMARY:
This study is being carried out in order to evaluate a new cancer vaccine called IMA970A combined with CV8102, a new adjuvant for the treatment of liver cancer (hepatocellular carcinoma). It will be investigated whether IMA970A and CV8102 is safe and can trigger an immune response against the tumor, which may prevent the tumor (cancer) from recurring or spreading or may even lead to tumor shrinkage following the standard treatments the patients have previously received.

DETAILED DESCRIPTION:
The trial is designed as a single-arm, open-label, multi-center, first-in-man phase I/II study investigating an off-the-shelf, multi-peptide-based HCC vaccine (IMA970A) plus CV8102 adjuvant (RNAdjuvant®) following a single pre-vaccination infusion of low-dose cyclophosphamide (CY) acting as an immunomodulator, in patients with very early, early and intermediate stage HCC.

The study treatment is applied without any concomitant anti-tumor therapy, with the intention to reduce the risk of tumor recurrence/progression in patients who have received all indicated standard treatments.

Overall, it is planned to treat about 40 patients with IMA970A (off-the-shelf vaccine) plus CV8102 (adjuvant) plus a single low-dose of pre-vaccination CY acting as an immunomodulator in the HepaVac-101 study.

Patients are requested to sign the 1st informed consent (IC 1) for screening 1 procedures (blood drawings for Human Leukocyte Antigen (HLA) typing and for cellular immunomonitoring, capture of demographics and staging of disease [routinely performed, older images may be used if requirements are met]), which takes up to 4 weeks. Thereafter, patients receive indicated standard treatment followed by recovery, which lasts for at least 4 weeks and up to 12 weeks. The main-phase with full safety surveillance starts with the patient's signature of the 2nd informed consent (IC 2) and lasts until the end of the EoV (End-of-Visit, Visit 10) Visit (4-6 weeks after last vaccination). For each patient this main-phase lasts up to approx. 6.5 months consisting of up to 4 weeks screening 2, about 4.5 months vaccination period and about 4 weeks follow up (until EOV Visit [Visit 10]).

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years
2. HLA type: HLA-A*02 and/or HLA-A*24 positive (Screening 1)
3. Very early, early and intermediate stage (Barcelona Clinic Liver Cancer (BCLC) stage 0, A, B disease) hepatocellular carcinoma (HCC) diagnosed by biopsy or resected tissue (pathohistological diagnosis) or imaging findings (non-invasive criteria) following any standard treatment (e.g. hepatic resection, Radiofrequency Ablation / Percutaneous Ethanol injection (RFA/PEI), Transarterial chemoembolization (TACE) and SIRT) and without any evidence of active disease that warrant further treatment

   1. Pathohistological diagnosis of HCC based on biopsy is required for all nodules occurring in non-cirrhotic livers, and for those cases with inconclusive or atypical imaging appearance in cirrhotic livers
   2. Non-invasive criteria can only be applied to cirrhotic patients and need to be based on imaging techniques obtained by 4-phase multi-detector CT scan or dynamic contrast-enhanced MRI and on the identification of the typical hallmark of HCC (hypervascular in the arterial phase with washout in the portal venous or delayed phase). One imaging technique is sufficient for nodules beyond 1 cm (> 1 cm) in diameter.
4. Patients for whom no standard anti-tumor therapy is indicated for the next 3 months (until after visit 7); thereafter any standard anti-tumor therapies applied for the treatment of BCLC stage 0, A and B HCC (e.g. RFA/PEI, TACE, and SIRT) are allowed to be applied in combination with the study treatment. Patients for whom treatment for advanced disease (e.g. sorafenib) is indicated will be withdrawn from study treatment.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0
6. Child-Pugh A5-6 and B7 disease or no liver function impairment
7. Able to understand the nature of the study and give written informed consent
8. Willingness and ability to comply with the study protocol for the duration of the study
9. Female patients who are post-menopausal (no menstrual period for a minimum of 1 year without any alternative medical cause), or surgically sterile (bilateral salpingectomy, bilateral oophorectomy, or hysterectomy) or practice a highly effective method of birth control from signing of IC 2 by the patient to visit 10/EoV or last study visit

   1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation applied intravaginal or transdermal for a minimum of 1 full cycle (based on the patient's usual menstrual cycle period) before first study drug application
   2. Progestogen-only hormonal contraception associated with inhibition of ovulation applied via injection or implant for a minimum of 1 full cycle (based on the patient's usual menstrual cycle period) before first study drug application
   3. Total abstinence from sexual intercourse is acceptable, if it was established prior to the trial and if this is the preferred and usual lifestyle of the patient.
   4. Intrauterine device (IUD) and intrauterine hormone-releasing system (IUS).
10. Male patients willing to use contraception (condoms with spermicidal jellies or cream) or have undergone bilateral orchiectomy and his non-pregnant WOCBP (women of childbearing potential partner) willing to use contraception (a highly effective method of birth control, see criteria above) from signing of IC 2 by the patient to visit 10/EOV or last study visit, however, at least 100 days after application of CY at Visit C

Exclusion Criteria:

1. Any prior systemic anti-tumor treatment (including drug or treatment regimen, approved or experimental) within 2 weeks before CY application
2. Concurrent participation in a clinical trial
3. Liver transplanted patients; patients who are on the liver transplantation waiting list are allowed to be enrolled
4. History of other malignancies within the last 3 years except for adequately treated except cervical carcinoma in situ, basal cell carcinoma and superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to signing of IC 2 by the patient
5. Patients with a history or evidence of systemic autoimmune disease, e.g. rheumatoid arthritis, multiple sclerosis, systemic lupus erythematodes (SLE), scleroderma, Sjögren's syndrome, Wegener's granulomatosis, Guillain-Barre syndrome
6. Need for concomitant treatment with immunosuppressive drugs or other immune-modifying drugs. The use of inhaled and nasally applied steroids, as well as topical steroids outside the vaccination area are permitted
7. Any medically diagnosed or suspected condition of immunodeficiency or medical history thereof
8. Known HIV infection
9. Any other known infection with a biological agent that can cause a severe disease and poses a severe danger to lab personnel working on patients' blood or tissue. Examples are: rabies, Mycobacterium leprae, Plasmodium falciparum, Coccidiodes immitis
10. Acute and active infections requiring oral or intravenous antibiotics, antiviral or antifungal therapy within 30 days prior to signing of the IC 2 by the patient (exception: Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infections; direct-acting antivirals may be applied as medically indicated.)
11. Patients undergoing renal dialysis or with relevant chronic renal failure
12. Abnormal laboratory values as specified below:

    1. Hematology: Hemoglobin (< 8.5 g/dl), platelets (< 75,000/µl), leukocytes (< 2,500/µl), neutrophils (< 1,000/µl), lymphocytes (< 500/µl)
    2. Liver function: serum bilirubin (≥ 3 x ULN), Alanine aminotransferase (ALAT) or Aspartate aminotransferase (ASAT) (≥ 5 x ULN)
    3. Renal function: serum creatinine (≥ 1.5 x ULN)
13. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics drugs)
14. Encephalopathy
15. Clinically relevant ascites with the only exception of patients that remain free from symptomatic ascites under low-dose diuretics (Spironolactone >100 mg daily and Furosemide >40 mg daily).
16. Hypersensitivity to the study drugs (CY, IMA970A, or CV8102) including excipients and to CT/MRI contrast agent
17. Known type I allergy to beta-lactam antibiotics
18. Evidence of current alcohol or drug abuse
19. Patient dependent on the sponsor or an investigator (e.g. employee, relative)
20. Serious intercurrent illness, which according to the investigator, poses an undue risk to the patient when participating in the trial, including, but not limited to, any of the following:

    1. Clinically significant cardiovascular disease (e.g., uncontrolled hypertension; clinically significant cardiac arrhythmia, clinically significant QT-prolongation),
    2. New York Heart Association class III-IV congestive heart failure,
    3. Symptomatic peripheral vascular disease,
    4. Severe pulmonary dysfunction,
    5. Psychiatric illness or known social situation that would preclude study compliance.
    6. Systemic inflammatory condition
21. Less than 6 months since any of the following:

    1. Myocardial infarction,
    2. Severe or unstable angina pectoris,
    3. Coronary or peripheral artery bypass graft,
    4. Cerebrovascular event incl. transient ischemic attack,
    5. Pulmonary embolism / deep vein thrombosis (DVT)
22. Patients with contra-indications for treatment with cyclophosphamide (acute infections, bone-marrow aplasia, urinary tract infection, acute urothelial toxicity from cytotoxic chemotherapy or radiation therapy, urinary outflow obstruction)
23. Pregnancy or breastfeeding
24. Any condition which in the judgment of the investigator would place the patient at undue risk or interfere with the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Through study completion, up to two years
  Safety assessments will consist of continuous monitoring and reporting of adverse events (AEs) including serious adverse events (SAEs), regular monitoring of vital signs, ECOG performance status and regular conduct of physical examinations and laboratory assessments (hematology, clinical [bio]chemistry including C reactive protein (CRP) and Glomerular Filtration rate (GFR), coagulation test, assessment of viral infection, thyroid function test (TFT), urinalysis), electrocardiogram (ECG) and pregnancy tests (if applicable). Additionally, an Independent Data Safety Monitoring Board (DSMB) will be implemented to evaluate safety data independently and at defined intervals.
Immunogenicity (T-cell response in peripheral blood) | Up to two years
  The assessment of immunogenicity will be performed for all patients using standardized immunomonitoring assays. Peripheral blood mononuclear cells (PBMCs) of patients will be analyzed for the occurrence of T-cell responses to peptides contained in IMA970A vaccine before application of standard therapy, such as before and after vaccination. The induction of immune responses by IMA970A vaccine will be subsequently analyzed.

SECONDARY OUTCOMES:
Additional immunological parameters in blood (e.g. regulatory T-cells, myeloid-derived suppressor cells) | Up to two years
  Analysis of other immune cell populations that may influence T-cell responses such as regulatory T cells (Tregs) and myeloid-derived suppressor cells (MDSC) (cellular biomarkers) will be performed using PBMCs
Infiltrating T-lymphocytes, immune cells and potential other (bio)markers in tumor tissue | Up to two years
  Analysis of paraffin-embedded tumor tissues (also potentially in liquid-nitrogen frozen tissue, if available) will be performed to characterize both the tumor cells and the tumor-infiltrating components by immunohistochemistry (IHC) and potentially other analysis techniques. Classical hematoxylin-eosin (HE) staining will be first performed to assess the cellular and stroma composition of the tumor tissue. Markers such as Cytokeratin 8, Cytokeratin 18 and HepPar-1, will be assessed to distinguish tumor cells from other cellular components. The tumor infiltrating cells will be characterized to assess leukocyte subpopulations such as myeloid (monocyte-macrophages, granulocytes) and lymphoid (T, B, NK) cells.
Assessment of the potential impact of the standard therapy on the natural imune response to peptides contained in IMA970A | Up to two years
  The assessment of the natural immune response to peptides contained in IMA970A will be performed before start of standard anti-tumor therapy and thereafter to assess whether the selected standard therapy has an influence on a potentially pre-existing (natural) immune response.
Time to progression (TTP) | Up to two years
  The time-related secondary efficacy endpoint for the trial is time-to-progression, with time being measured from baseline CT/MRI scan (at Visit B) to documented tumor progression.
Overall survival (OS) | Patients will be followed for overall survival every 2 months for up to 3 years, after having completed the interventional part of the study at EOV/Visit 10.
  Patients will be followed for overall survival

CONTACTS AND LOCATIONS:
Locations (6):
- Universitair Ziekenhuis Antwerpen (UZA), Division of Gastroenterology and Hepatology, Edegem, Belgium
- Universitätsklinik für Allgemeine, Viszeral- und Transplantationschirurgie, Tübingen, Germany
- Italy (2):
  - Istituto Nazionale Tumori "Pascale" (INTNA), Napoli
  - Ospedale Sacro Cuore-Don Calabria U.O.C. Oncologica Medica, Negrar
- Universidad de Navarra (NAVAR), Internal Medicine, Pamplona, Spain
- The University of Birmingham, School of Immunity and Infection, College of Medical and Dental Science (BHAM), Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loffler MW, Gori S, Izzo F, Mayer-Mokler A, Ascierto PA, Konigsrainer A, Ma YT, Sangro B, Francque S, Vonghia L, Inno A, Avallone A, Ludwig J, Alcoba DD, Flohr C, Aslan K, Mendrzyk R, Schuster H, Borrelli M, Valmori D, Chaumette T, Heidenreich R, Gouttefangeas C, Forlani G, Tagliamonte M, Fusco C, Penta R, Inarrairaegui M, Gnad-Vogt U, Reinhardt C, Weinschenk T, Accolla RS, Singh-Jasuja H, Rammensee HG, Buonaguro L. Phase I/II Multicenter Trial of a Novel Therapeutic Cancer Vaccine, HepaVac-101, for Hepatocellular Carcinoma. Clin Cancer Res. 2022 Jun 13;28(12):2555-2566. doi: 10.1158/1078-0432.CCR-21-4424. PMID 35421231